CLINICAL TRIAL: NCT04006535
Title: Identification of Susceptibility Loci and Genes for Systemic Vasculitis Risk, by Analyzing Whole Exome Sequencing of Familial and Pediatric Forms of Vasculitis (FAMILYVASC Study)
Brief Title: Whole Exome Sequencing of Familial and Pediatric Forms of Vasculitis
Acronym: FAMILYVASC
Status: Recruiting | Type: Observational
Sponsor: Benjamin Terrier (Other)
Responsible Party: Sponsor-Investigator, Benjamin Terrier, Professor, French Vasculitis Study Group
Organization: French Vasculitis Study Group (Other)
Other Study IDs: 2019-A00188-49
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Vasculitis
Keywords: Vasculitis
MeSH Terms: conditions — Vasculitis | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples will be collected for genetic analysis and identification of susceptibility loci and genes for the risk of vasculitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: genetic analysis — Saliva sample collection for genetic analysis

SUMMARY:
The FAMILYVASC study is a prospective observational study which will aim to identify susceptibility loci and genes for systemic vasculitis risk in patients with familial or pediatric forms of vasculitis. Genetic analysis based on whole exome sequencing will be carried out through salivary DNA.

ELIGIBILITY:
Inclusion criteria for subjects with vasculitis

* Children and adults
* Patients with vasculitis, as defined in the Chapel Hill International Classification in its revised version of 2012
* Patient information and signed informed consent
* Pregnant and breastfeeding women can be included in the study

Inclusion criteria for healthy subjects

* Children and adults
* Do not have vasculitis, as defined in the Chapel Hill International Classification in its revised version of 2012, or relatives on the 1st; 2nd; 3rd or 4th degree of a patient with vasculitis
* Patient information and signed informed consent
* Pregnant and breastfeeding women can be included in the study

Exclusion criteria:

* Refusal of consent or inability to obtain consent
* Dementia or unauthorized patient, for psychiatric or intellectual failure reasons, to receive information about the protocol and to give informed consent.
* Uncooperative patient, or any pathology that could make the patient potentially non-compliant to the study procedures, and patients interned for regulatory or legal reasons.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult and childhood patients (no age limit) with familial and pediatric forms of vasculitis as defined in Chapel Hill's international nomenclature in its revised 2012 version.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of susceptibility loci and genes | At the moment of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Terrier, MD, PhD, Principal Investigator — French Vasculitis Study Group
Locations (1):
- Hôpital Cochin - Department of Internal Medicine, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.vascularites.org